CLINICAL TRIAL: NCT03708965
Title: An Extension Study of JR-141-BR21 in Patients With Mucopolysaccharidosis II
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: JCR Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JR-141-BR22
Record Dates: First submitted 2018-09-27; First posted 2018-10-17 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Mucopolysaccharidosis II
MeSH Terms: conditions — Mucopolysaccharidosis II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- JR-141 (Experimental): Subjects will be assigned to 1.0, 2.0 or 4.0 mg of JR-141 per kg of body weight once every week (the same dose taken during the previous study) in the beginning of the study.
  During the study, the dose of all subjects will be switched to the selected one*.
  * The dose was determined to be 2.0 mg/kg/week based on the safety and efficacy data of JR-141-BR21 study.
  Interventions: Drug: JR-141

INTERVENTIONS:
Drug: JR-141 — IV infusion (lyophilized powder)

SUMMARY:
A Phase II open-label, parallel group, 2 sites (Brazil), designed to evaluate the long term safety and efficacy of study drug for the treatment of the MPS II.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will have completed clinical trial JR-141-BR21.
* Capable of providing written consent by himself, unless the patient is under the age of 18 years at the time of informed consent process, or it is not possible to obtain consent from the patient himself due to his intellectual disabilities associated with MPS II.
* In the case of a patient who is under the age of 18 years or from whom it is not possible to obtain consent due to his intellectual disabilities associated with MSP II, he may be included if written consent can be provided by legal representative; however written consent should be obtained from the patient himself too, wherever possible.

Exclusion Criteria:

* Refusal to sign the informed consent form.
* Unable to perform the study procedures, except for neurocognitive testing.
* Previous engrafted BMT/HSCT.
* Judged by the investigator or subinvestigator as being unable to undergo lumbar puncture, including those who have difficulties in taking a position for lumber puncture due to joint contracture or those who are likely to experience difficulty breathing during the lumbar puncture process.
* Judged by the investigator or subinvestigator to be ineligible to participate in the study due to a history of a serious drug allergy or sensitivity.
* Otherwise judged by the investigator or subinvestigator to be ineligible to participate in the study out of consideration for the subject safety.

Min Age: 0 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | From screening up to the end of study, up to approximately 5 years

SECONDARY OUTCOMES:
Urinary heparan sulfate concentrations | through study completion, an average of 52 weeks, up to approximately 5 years
Urinary dermatan sulfate concentrations | through study completion, an average of 52 weeks, up to approximately 5 years
Serum heparan sulfate concentrations | through study completion, an average of 52 weeks, up to approximately 5 years
Serum dermatan sulfate concentrations | through study completion, an average of 52 weeks, up to approximately 5 years
Liver and spleen volumes (MRI) | through study completion, an average of 52 weeks, up to approximately 5 years
Echocardiography | through study completion, an average of 52 weeks, up to approximately 5 years

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Grupo de Pesquisa Clínica em Genética Médica - HCPA, Porto Alegre
  - Igeim - Unifesp, São Paulo

IPD SHARING:
Plan to Share IPD: No